# Clinical Investigation Plan

# **CP300**

Assessment of new enhanced ostomy device in real-life settings in subjects having a stoma

November 2018 – March 2019

Master

This confidential document is the property of Coloplast A/S. No unpublished information contained herein may be disclosed without written approval of Coloplast A/S.





<sup>&</sup>lt;sup>1</sup> Attachment composed by The Danish National Committee on Health Research Ethics, about subject's rights in a clinical investigation.

| VERSION<br>NUMBER | ISSUED BY<br>(INITIALS) | COMMENTS (MAJOR CHANGES | SINCE LAST REVISION) |
|---|---|---|---|

# > TABLE OF CONTENTS

| 1. | List of personnel involved in the Investigation | 9 |
|---|---|---|
| 1.1. | . Sponsor representatives | 9 |
| 1.2 | . Investigators | 9 |
| 1.3 | . Other | 10 |
| 2. | Identification and description of the investigational device | 11 |
| 2.1. | . Manufacture | 11 |
| 2.2 | . Description of investigational device | 11 |
| 2.3 | . Identification, traceability and labelling of device | 11 |
| 2.4 | . Clinical investigation intended use of device | 12 |
| 2.5 | . Intended population for the device | 12 |
| 2.6 | . Handling and training | 12 |
| 2.7 | . Comparator product(s) | 13 |
| 3. | Justification for the conduct of the clinical investigation | 14 |
| 4. | Investigational device and clinical investigation risks and benefits | 15 |
| 4.1. | . Anticipated clinical benefits | 15 |
| 4.2 | . Anticipated risks and disadvantages | 15 |
| 4.3 | . Benefits versus risks | 16 |
| <i>5.</i> | Aim, objectives and hypotheses of the clinical investigation | 17 |
| 5.1. | . Aim | 17 |
| 5.2 | . Objective | 17 |
| 5.3 | . Hypotheses | 17 |
| 6. | Design of the clinical investigation | 18 |
| 6.1 | . General | 18 |
| 6.2 | . Investigational device and comparator(s) | 27 |
| 6.3 | . Subjects | 27 |
| 6.4 | . Procedures | 31 |
| 6.5 | . Supplementary material and equipment | 40 |
| 6.6 | . Monitoring Plan | 40 |
| 7. | Statistical considerations | 43 |
| 7.1 | . Statistical design, method and analytical procedures | 43 |
| 7.2 | . Sample size | 44 |
| 7.3 | . Level of significance and power | 45 |
| 7.4 | . Drop-out | 45 |
| 7.5 | . Pass/fail criteria | 45 |

| 7.6 | i. lı | nterim analysis | 45 |
|---|---|---|---|
| 7.7 | '. S | Statistical reason for termination of investigation | 45 |
| 7.8 | 3. C | Deviation(s) from statistical plan | 46 |
| 8. | Da | ta managementta | 46 |
| 8.1 | . С | oata review, database cleaning, and issuing and resolving data queries | 46 |
| 8.2 | 2. V | erification, validation and securing of electronic clinical data systems | 46 |
| 8.3 | 3. C | Pata retention | 46 |
| 9. | An | nendments to the CIP | 47 |
| 10. | Cli | nical Investigation Plan deviations | 48 |
| 10 | .1. | Deviations | 48 |
| 10 | .2. | Violations | 48 |
| 11. | De | vice Accountability | 49 |
| 12. | Sta | atement of compliance | 50 |
| 12 | .1. | Ethics committee and regulatory authorities | 50 |
| 12 | .2. | Data protection | 50 |
| 12 | .3. | Indemnity | 51 |
| 12 | .4. | Financial conditions | 51 |
| 13. | Inf | ormed consent process | 51 |
| 14. | Ad | verse events, serious adverse events and device deficiencies | 53 |
| 14 | .1. | Adverse events | 53 |
| 14 | .2. | Device deficiency | 54 |
| 14 | .3. | Serious adverse events | 54 |
| 14. | .4. | Medical care of subjects | 55 |
| 14. | .5. | Reporting and timelines | 55 |
| 15. | Su | spension or premature termination of the clinical investigation | 57 |
| 16. | Cli | nical investigation report | 58 |
| 17. | Pu | blication policyblication policy | 59 |
| 17. | .1. | General | 59 |
| 18. | Bil | bliography | 60 |
| 20. | Ap | pendix | 61 |
| 20 | .1. | Appendix 1: LOCAL CHANGE LOG | 61 |
| 20 | .2. | Appendix 2: Leakage scale questionnaire | 62 |
| 20 | .3. | Appendix 3: Quality of life questionnaire | 64 |
| 20 | .4. | Appendix 4: Safety Interview guide | 66 |
| 20 | .5. | Appendix 5: Interview guide (V6) and Follow-up | 67 |

#### SYNOPSIS OF THE CLINICAL INVESTIGATION

#### Aim and Objective

The aim of the investigation is to investigate the performance of a baseplate

The **primary objective** is to investigate whether a new baseplate

The secondary objective is to investigate the safety of a new baseplate

#### Primary endpoint and explorative endpoint(s)

Primary endpoint: Trans epidermal water loss (inner circle around stoma).



#### Pass/fail criteria

No formal success criteria are applied in this explorative investigation. The investigation will provide valuable insight into how the peristomal skin reacts

#### Design of the investigation

This investigation is a controlled, comparative, multicentre investigation, that consist of two test periods. During Test Period 1 the subjects will be asked to use SenSura® Mio (Comparator) for baseline data for 14 (-2/+15) days. Hereafter they will be asked to use the test product for 28 (-4/+12) days during Test Period 2.

Before the test periods the subjects are invited for an inclusion visit (V0). Subjects sign all consent forms at this visit before continuing the investigation. Hereafter, the subjects will complete five test visits (V1, V2, V4, V5 and V6) and one safety visit at site (V3). After termination, a follow-up visit may be conducted at the subject's home.

### **Population**

The population in this investigation includes 25 subjects with an ileostomy or a colostomy with liquid output that comply with the following in- and exclusion criteria:

| Inclusion criteria To be included the subjects must: | Exclusion criteria The subjects are not allowed to participate in case they: |
|---|---|
| Have given written informed consent | Are currently receiving or have within the past two months re-<br>ceived radio-and/or chemotherapy (low doses chemotherapy<br>are allowed for other indications than cancer, e.g. below 15 mg<br>methotrexate for rheumatoid arthritis) |

| Have an ileostomy or a colostomy with liquid* output (as their usual output) * Bristol Scale: 6-7 | Are currently receiving or have within the past month received topical steroid treatment in the peristomal skin area (e.g. lotion or spray) or systemic treatment* (e.g. injection or tablets). *Investigator will decide on case basis whether the treatment is accepted under the protocol |
|---|---|
| Be at least 18 years of age and have full legal capacity | Get a positive result of a pregnancy test for women of childbearing age/fertile (**clarified in section 6.3.2) |
| Have had their stoma for at least three months | Are breast feeding |
| Be able to use products with max cut size 45 mm | Are participating in other interventional clinical investigations or have previously participated in this investigation Exception: Participation in other Coloplast in-house clinical investigations is accepted under the circumstances that the subject has paused the activities in the investigation and are otherwise complying with the inclusion and exclusion criteria of this (CP300) protocol. |
| Have self-reported problems with leakage** (three times within 14 days) **Leakage: Leakage is defined as output from the stoma on the backside of the baseplate (underneath the baseplate) | Have known hypersensitivity towards any of the products used in the investigation |
| Use a flat SenSura® Mio or a flat SenSura® with standard adhesive as their current product Standard adhesive: Not extended wear adhesive | |
| Minimum change of baseplate at least once every 3 <sup>rd</sup> day | |
| Are willing and suitable (determined by investigator/study nurse) to use the test product and comparator without using a paste/mouldable ring during the investigation | |
| Are willing and suitable (determined by investigator/study nurse) to use a 1-piece product during the investigation | |

# **Test products**

The test product is a non-CE marked stoma product with flat custom cut adhesive, with open maxi bags and with the intended use of collecting output from a stoma. The product is based on the SenSura® Mio 1-piece stoma product (already CE-marked and launched),

The comparator product is the SenSura® Mio 1-piece stoma product.

# Investigation approval

The investigation will be approved by the Ethical committees and the competent authorities in the participating countries before investigation initiation.

# > SIGNATURE PAGE

All parties declare by their signature on the electronic or the separate signature page to follow the Clinical Investigation Plan CP300 in accordance with the Declaration of Helsinki, ISO 14155 and the Medical Device Directive/Medical Device Regulation.

# 1. List of personnel involved in the Investigation



In case of emergency, please contact the Coordinating Clinical Manager from the above list of sponsor representatives.

# 1.2. Investigators

The Coordinating Clinical Manager is responsible for maintaining an updated Site Personnel Contact Details list of all Principal Investigators, investigation sites and institutions. Details of all Principal Investigators, investigators, including a CV, are maintained in the Sponsor File.

Qualified site personnel can perform investigation related tasks as investigator representatives. This delegation will be documented in the "Site Personal Signature and Delegation List" for each site. All investigators and investigator representatives will receive oral and written training in all investigation related tasks before they can begin any investigation related tasks. The training will be documented in the Clinical Investigation Training Log at each site.

#### 1.3. Other

CROs may be used to help conduct the investigation as Sponsor representatives in one or more countries. The CROs, their role and responsibilities will be listed in the Site Personnel Contact Details list.

## 2. Identification and description of the investigational device

The test product is a non-CE marked stoma product with flat custom cut adhesive, with open maxi bags and with the intended use of collecting output from a stoma. The product is based on the SenSura® Mio 1-piece stoma product (already CE-marked and

#### 2.1. Manufacture

Coloplast A/S, Holtedam 1-3, 3050 Humlebæk, Denmark, manufactures the investigational device.

# 2.2. Description of investigational device



#### 2.3. Identification, traceability and labelling of device

The products will be packed in retail boxes with ten 1-piece products in each box. Labelling of the test products (1-piece) is shown in the figure below. These labels will be attached to the retail boxes.

Table 1: Illustration of labels for the test product for 1-piece devices. Lot number and expiry date will be added before release of products.



# 2.4. Clinical investigation intended use of device

The ostomy bag is intended to collect output from a stoma. The adhesive is intended to fix the bag and adhere to intact peristomal skin around the stoma.

#### 2.5. Intended population for the device

The intended population for the device is people with an ileostomy or a colostomy with liquid output.

#### 2.6. Handling and training

The handling of the test products is described in details in the Instruction for Use (IFU), which is included in all boxes with test products. It is stated in the IFU that the test products are for single-use and must be stored horizontally under dry and not freezing conditions, and should be kept away from direct sunlight. Reprocessing, washing, disinfection, and sterilisation may compromise product characteristics, causing additional risk of physical harm to or infection of the user<sup>2</sup>.

<sup>&</sup>lt;sup>2</sup> Product Risk Management Report – Clinical Study CP300 Genesis (VV0227119)

All Investigators / investigator representatives will receive training by sponsor / investigator in the handling and correct use of the test products. The Investigator/investigator representative will train the subjects in the correct use of the test products.

# 2.7. Comparator product(s)

As the comparator product is already on the market and will be used within the intended use in this clinical investigation, it is not considered an investigational device according to ISO 14155:2011 and is thus not described here. Please refer to the ISO 14155:2011 for details.

# 3. Justification for the conduct of the clinical investigation

| People with abdominal stomas (especially ileostomis | sts) have, despite development of better stoma products, |
|---|---|
| problems with leakage | influence quality of life negatively [2]. To overcome this, |
| Coloplast A/S has developed a new stoma product v | with a baseplate |
| The aim is to seek knowledge of whe | ther the new baseplate can protect the skin |

# 4. Investigational device and clinical investigation risks and benefits

The clinical investigation is conducted in accordance with current law and applicable standards (see section 12). The rights, safety and well-being of the subjects shall prevail over science and society. All investigators and investigator representatives will be instructed in performing their job with conscientiousness and care.

#### 4.1. Anticipated clinical benefits



#### 4.2. Anticipated risks and disadvantages

#### **Anticipated risks**

A number of risks connected to use of the test product have been identified in the Product Risk Assessment. All risks will be mitigated before release of products for the clinical investigation. The risk management process has been performed in accordance with the requirements stated in ISO 14971:2012 and in accordance with internal Coloplast procedures, including design verification, validated test methods, risk analysis and completion of a biological report for the test product.

The following risks will also be mitigated by actions during the clinical investigation, specified in this Clinical Investigation Plan:

Irritated skin (intact or non-intact): Use of the product can lead to intact or non-intact irritated skin. To mitigate and reduce the risk, the users will be trained, according to the IFU, in preparation of the product (e.g. hole size), preparation of skin before application (e.g. cleaning and wiping), application of product (e.g. correct position and applying pressure to the baseplate), removal of product and storage of the product.



#### Residual risks

Residual risks will be assessed after mitigation of the risks.

#### Disadvantages

Disadvantages during the investigation could be the extra workload related to completion of questionnaires, visits at site and using the clinical app at each change of product.

Danish Competent Authorities registration number: 2017102759 and CIV-ID: CIV-17-10-02-021866

<sup>&</sup>lt;sup>3</sup> Danish Ethical Committee registration number: H-17031767

#### Interactions with concomitant medication

There is no known interaction between the use of the stoma products used in the clinical investigation and concomitant medication.

#### 4.3. Benefits versus risks

The participating subjects will contribute with important information for development of new stoma products, that may have less negative impact om the peristomal skin. Due to the actions taken to mitigate the above-mentioned risks, the risks and disadvantages when participating in this clinical investigation are estimated as low. The subject's heath will not benefit directly from this investigation but they may benefit from the use of the new stoma product through less irritated peristomal skin and improved quality of life and in the future.

# 5. Aim, objectives and hypotheses of the clinical investigation

#### 5.1. Aim

The aim of the investigation is to investigate the performance of a baseplate with a

# 5.2. Objective

The **primary objective** is to investigate whether a new baseplate

The secondary objective is to investigate the safety

# 5.3. Hypotheses

The hypothesis is that investigation is explorative, there is no formal criteria for success.

# 6. Design of the clinical investigation

#### 6.1. General

This investigation is a controlled, comparative, multicentre investigation, that consist of two test periods. During Test Period 1 the subjects will be asked to use SenSura® Mio (Comparator) for baseline data for 14 (-2/+15) days. Hereafter the subjects will be asked to use the test product for 28 (-4/+12) days during Test Period 2. During the test periods the subjects can change their product as often as needed, but at least every third day.

Before the test periods the subjects are invited for an inclusion visit (V0). Subjects sign all consent forms at this visit before continuing the investigation. Hereafter, the subjects will complete five test visits (V1, V2, V4, V5 and V6) and one safety visit at site (V3). After termination, a follow-up visit may be conducted at the subject's home.

Biological materials (faeces) will be collected during the investigation for analysis only related to this investigation. Therefore, an Investigational BioBank will be created for this purpose. The samples of biological materials will be stored in a separately CP300 allocated freezer at site, and send on an ongoing basis to Coloplast A/S, Humlebæk, Denmark. The samples of biological materials will not be stored longer than it takes to collect and analyse the samples. The sample will be destroyed directly after analysis. The Biobank will be closed when all output samples have been analysed and destroyed, or at three months after last patient out.

Please see section 6.4.1 Clinical Investigation-related Procedure for more information about procedures during the investigation.

# 6.1.1. Endpoints

Table 2: List of Primary, Explorative and Safety Endpoints. <sup>1</sup>Investigator can delegate the task to trained site personnel. <sup>2</sup>Only completed by subject at the first 14 change of products during test period 1 and completed by subject at every change of product during test period 2.

| | Endpoint | Type of assessment | Assessed<br>by | V1 | V2 | V3 | V4 | V5 | V6 | Product change |
|---|---|---|---|---|---|---|---|---|---|---|
| Primary end-<br>point | Trans Epidermal Water Loss (TEWL) • Inner circle | Objective skin measurement<br>[TEWL] = gm <sup>-2</sup> h <sup>-1</sup> | Investigator <sup>1</sup> | X | X | | X | Х | X | |
| Explorative | | | | | | | | | | |
| | | | | | 14 pp 40 | | | | | |
| | | | | | V <sub>F</sub> N | | | | | |
| | | | S. Se | | P <sub>12</sub> is | | | | | |







| Endp | point | Type of assessment | Assessed<br>by | V1 | | V3 | V4 | V5 | V6 | Product change |
|---|---|---|---|---|---|---|---|---|---|---|
| - | | | | | | | I | ı | | |
| | | | | | | | | I | | |
| 2 | | | | | | | | | | |
| | | 120 | | | - | - | e. <b>■</b> | | | |

# 6.1.2. Qualitative data

| Qualitative data | Type pf assessment |
|------------------|--------------------|

# 6.1.3. Baseline data

Registered at the inclusion visit (V0) by Investigator or a delegate hereof

- Date of informed consent (date)
- Date of visit (date)
- Check of inclusion criteria
- Check of exclusion criteria
- Subject number (number)

#### Demographic

- Date of birth (date)
- Gender (male/female)
- Height (number cm)
- Weight (number kg)

#### Stoma

- Age of stoma (year when created)
- Type of stoma (ileostomy/colostomy)
- Cause of the stoma (Crohn's disease/Colitis ulcerosa/ Cancer/ Other)
- Size of the stoma (diameter on widest place and height)
- Shape of the stoma (round/oval/irregular)
- Does your stoma change colour? (Yes/No)
  - If yes, please describe
- Does your stoma sometimes secrete excessively (weeping stoma)? (Yes/No)
  - If yes, please describe?
- Does your stoma change shape (change in diameter, change in length)? (Yes/No)
  - If yes, please describe?
- Does your stoma bleed regularly? (Yes/No)
  - If yes, please describe?
- Does your stoma change behaviour due to?
  - exercise? (Yes/No)
    - if yes, please describe
  - specific foods? (Yes/No)
    - if yes, please describe
  - hydration level? (Yes/No)
    - if yes, please describe
  - Other? (Yes/No)
    - If yes, please describe

#### Current product

- What is your Current product (brand, product name, item number, size, product type (1-piece)
- Are you used to cut the baseplate? (Yes/No)
  - If yes, how much is cut off from the baseplate (template of the baseplate where the cut is drawn upon, max cut in mm)?

#### Peristomal skin area

- How often do skin complications occur? (Daily, Every 2-3 days, Once a week, Once every second week, More rarely)
- Body profile with body check tool

#### Leakage/output

What is the frequency of your output? (All the time (continuous)/with regular intervals/with irregular intervals)

#### 6.1.4. Rationale for selection and measurement of endpoints

The primary endpoint, TEWL, is a standardised non-invasive method for describing the barrier function of the skin. Damage to the skin surface will lower the barrier of the skin and thereby increase the water loss. This measurement is therefore used as primary endpoin

Additional skin measurements, assessments and the skin condition endpoints are all parameters describing the skin. Therefore, these are also essential to investigate if the new baseplate

The median wear time per subject in each period is used as endpoint, as it is considered a robust estimation of wear time.

Adverse events, device deficiencies, concomitant medication and safety questions comprise safety parameters. Qualitative interviews will give a subjective insight in the subject experience with the test product.

#### 6.1.5. Discussion of clinical investigation design

The new test product is intended for people with an ileostomy and for colostomists with liquid output. The two groups experience the same issues regarding leakage and skin problems and could therefore benefit from the product.

SenSura® Mio and SenSura® users are chosen and will be considered as one group, since results from a previous investigation<sup>4</sup> showed no difference between the two user groups regarding inner circle TEWL (primary endpoint).

The duration of Test Period 1 (14 (-2/+15) days) and two test visits in the period is found adequate to assess baseline data on the wear time, leakage pattern and skin condition of the subject. The test product is tested for 28 (-4/+12) days to ensure that the skin will have time to adjust to the new conditions, reach a steady state, and for the subjects to test an adequate number of products to give a thorough evaluation of the products.

To follow safety closely and ensure proper compliance and no unexpected events related to the test product, the first five subjects will be enrolled at the Coloplast Humlebæk Site DK001 (Sponsor). In addition, and due to Christmas holiday, follow-up logistics and planning purpose, the following subjects, at other sites than DK001, will be invited for the test visit 1 during week 49-51 (December 2018) and for their test visit 2 during week 1 and 2 (January 2019).

3

<sup>&</sup>lt;sup>4</sup> CP275 – A clinical investigation evaluating three new 1-piece ostomy products Danish Ethical Committee registration number H-17005054/Danish Competent Authorities registration number DMA-2017022387

In this investigation, a part of the information about the products is obtained via interviews (qualitative data). The interviews allow for detailed questions (in the form why, when, how) that can be adjusted individually per each subject's experience. This gives more details about the subject's experience with the test product. However, some drawbacks also occur with this method of obtaining information, as the interview data is subjective and cannot be quantified. The interviews may also cause a positive bias towards Coloplast. Thus, in this explorative investigation, the main endpoints are obtained by CRFs (from all subjects) and the interviews are used for supplementary information. The data collected by interviews will be handled confidentially, as all other data collected in this investigation.

The investigation is not blinded because the test product and SenSura® Mio are visible different from each other. If the subjects have a preconceived attitude to the test products or SenSura® Mio bias could occur for all subjective parameters.

# 6.2. Investigational device and comparator(s)

Subjects using 1-piece open products are expected to change their products every day. Therefore, they are expected to use 14 (-2/+15) of the comparator products during Test Period 1 and 28 (-4/+12) of the test products during Test Period 2.

To take the variety of visit windows, change patterns and distribution logistics to sites in different countries into account, a safety margin of products has been added. Therefore, the total number of products for this investigation is 2000 1-piece products.

The test product is based on the SenSura® Mio 1-piece products already on the market. Therefore, the comparator in this investigation is:

- 1-piece
  - SenSura® Mio 1-piece open, flat, maxi, neutral grey, 10-55 mm and circle filter

#### 6.3. Subjects

To be included in the investigation, the subjects must comply with the selection criteria described in section 6.3.1 and must not comply with the exclusion criteria described in section 6.3.2.

#### 6.3.1. Inclusion criteria for subject selection

Subjects interested in participating the clinical investigation must comply with the following criteria:

| Inclusion criteria To be included the subjects must: | Justification To ensure that: |
|---|---|
| Have given written informed consent | the subject participates voluntarily |
| Have an ileostomy or a colostomy with liquid* output (as their usual output) * Bristol Scale: 6-7 | only subjects which the product is aimed for will be included |
| Be at least 18 years of age and have full legal capacity | <ul> <li>the subject is competent and that data quality is<br/>high</li> </ul> |

| Have had their stoma for at least three months | <ul> <li>the initial post-operative problems are overcome,<br/>and that the subject is used to having an ostomy as<br/>well as changing the product before entering the<br/>investigation</li> </ul> |
|---|---|
| Be able to use products with max cut size 45 mm | |
| Have self-reported problems with leakage** (three times within 14 days) **Leakage: Leakage is defined as output from the stoma on the backside of the baseplate/underneath the baseplate | a potential change in leakage performance and<br>skin condition can be observed |
| Handle the Clinical App, test product and comparator product themselves | <ul> <li>the subject can take pictures and complete the<br/>CRF questions in the app, in addition to handle the<br/>products</li> </ul> |
| Use a flat SenSura® Mio or a flat SenSura® with standard adhesive as their current product Standard adhesive: Not extended wear adhesive | <ul> <li>the subjects will use a product with the same wear<br/>time</li> </ul> |
| Minimum change of baseplate at least once every 3 <sup>rd</sup> day | <ul> <li>To ensure that subjects change the products suffi-<br/>cient times during the investigation</li> </ul> |
| Are willing and suitable (determined by investiga-<br>tor/study nurse) to use the test product and com-<br>parator without using a paste/mouldable ring dur-<br>ing the investigation | a potential effect of the new baseplate cannot be detected |
| Are willing and suitable (determined by investiga-<br>tor/study nurse) to use a 1-piece product during the<br>investigation | <ul> <li>to ensure compliance to the protocol during the investigation</li> </ul> |

# 6.3.2. Exclusion criteria for subject selection

Subjects complying with the following criteria must be excluded from participation in the clinical investigation:

| Exclusion criteria The subjects are not allowed to participate in case they: | Justification |
|---|---|
| Are currently receiving or have within the past two months received radio-and/or chemotherapy (low doses chemotherapy are allowed for other indications than cancer, e.g. below 15 mg methotrexate for rheumatoid arthritis) | The skin undergoes major changes because of radio-<br>and/or chemotherapy, and as a consequence, the skin<br>might be more fragile to product changes. |
| Are currently receiving or have within the past month received topical steroid treatment in the peristomal skin area (e.g. lotion or spray) or systemic treatment* (e.g. injection or tablets). *Investigator will decide on case basis whether the treatment is accepted under the protocol | Steroid product on peristomal skin may interfere with<br>the skin condition. Use of steroid product can make<br>the skin more fragile to baseplate change. |
| Get a positive result of a pregnancy test for women of childbearing age/fertile** | Even though the ingredients and the recipes have been approved for humans, their effect on embryos, foetuses, and infants are unknown. |

| Are breast feeding | Even though the ingredients and the recipes have been approved for humans, their effect on embryos, foetuses, and infants are unknown. |
|---|---|
| Are participating in other interventional clinical investigations or have previously participated in this investigation Exception: Participation in other Coloplast in-house clinical investigations is accepted under the circumstances that the subject has paused the activities in the investigation and are otherwise complying with the inclusion and exclusion criteria of this (CP300) protocol. | Other interventional investigation guidelines/products may interfere with these investigational endpoints. Some of the Coloplast studies are taking place over a two-year period, where the subjects will be paused for longer periods between the visits - therefore they can participate in other Coloplast studies meanwhile. |
| Have known hypersensitivity towards any of the products used in the investigation | It is not ethical to include persons that know they are allergic to the products used in the investigation and it would also create bias, as these persons would give the product they are allergic to a more negative rating and most likely also create an AE. |

<sup>\*\*</sup> Besides a negative pregnancy test the women must also sign a document claiming that they will use safe contraceptives during the study period (i.e. contraceptive coil, hormone base contraceptives or surgical sterilisation). However, in some cases when the women are older than 50 years, but are not yet post-menopausal, the investigator may evaluate that it is not reasonable to ask these women to start using safe contraceptives for the duration of the investigation (e.g. if the subject is abstinent, the partner is surgically sterilised, or either subject or partner is infertile). In these cases, the investigator can include the women, but has a responsibility of ensuring that he/she has done what he/she can to prevent these subjects from becoming pregnant. As a minimum investigator, must talk to the women about the risk of and how to avoid unwanted pregnancy at inclusion.

#### 6.3.3. Recruitment and enrolment

The recruitment of potential subjects will commence only once authorisation has been received from the Regulatory Authorities and the EC.

Table 3: Table showing an overview of the recruitment process

| Recruitment<br>method | Coloplast Database | Advertisement | Patient records |
|---|---|---|---|
| Potential subjects | Recruitment will go through Coloplast own subject data- base (stoma care users) in Denmark and Sweden. Potential subjects are identi- fied by the following search- ing criteria in the Coloplast database: Has an ileostomy or co- lostomy 1-piece or unspecified Open or unspecified | Advertisement i.e. in local shops, sports facilities, local newspapers, social media and ostomy associations. The advertisement will state the contact information of relevant investigator(s) to contact. A CRO may help by receiving reply letters/mails and/or answering the phone from interested subjects. | Recruitment from hospitals, home care nurses and outpatient ostomy clinics will be via patient visit or screening of subject records kept at the participating sites. |

| | Be at least 18 years of | | |
|---|---|---|---|
| <b></b> | age | | T : |
| First contact | The identified potential sub- | Interested subject contact | The identified potential sub- |
| | jects will as first contact be | the investigator. | jects will be contacted and in- |
| | sent an Invitation and Reply | | formed about the investigation |
| | Letter by mail or email. | | by the investigator (via tele- |
| | If a potential subject does | | phone, letter or e-mail). |
| | not return the reply letter or | | |
| | answer the email, they may | | |
| | be contacted by phone, mail | | |
| | or email to make sure that | | |
| | they have received the ap- | | |
| | proach. | | |
| Second contact | If potential subjects return the | Reply Letter/reply to the email, o | or have called the investigator as |
| | first contact and are interested | , the Investigator or delegated s | ite personnel will contact the |
| | subjects by phone and give a s | short introduction to the investiga | ation and go over the inclusion |
| | and exclusion criteria. | | |
| | If the subjects do not meet the inclusion criteria or meet the exclusion criteria, this will be regis- | | |
| | tered at the Subject Screening | Log. | |
| Subject Infor- | If subjects are eligible and inte | rested in participating, then writt | en information about the investi- |
| mation Form | gation (subject information) wil | I be sent to the subjects to ensu | re that they are given the oppor- |
| | tunity to read about the investi | gation before a possible informa | tional visit, and so that they can |
| | prepare any possible questions | s they may have. The subject in | formation provides information to |
| | subjects about how to contact | the investigator or a representat | ive thereof, or a representative |
| | of the sponsor (name, telephor | ne number and e-mail address), | if they wish to learn more about |
| | the study. | | |
| First visit | If an eligible subject is interest | ed in participating after the first o | contact, a visit will be arranged in |
| Information visit | a room reserved to ensure priv | acy and quiet surroundings at th | ne investigators clinic/depart- |
| | ment. When arranging the visit | , it will be ensured, that the subj | ect has received the Information |
| | Form prior to the visit. The sub | jects will receive both written an | d verbal information about the |
| | I | nion to the informational visit an | |
| | visits. | | |
| | See section 13 for information | to be given to the subjects, as w | vell as the informed consent pro- |
| | cess. | , , | • |
| Enrolment and in- | The subjects have the right to | wait 24h before deciding on part | cicipation. If/when the subject de- |
| clusion visit (V0) | | | rms (see section 13). If a subject |
| ` ' | | t it is understood what the inves | , , |
| | 30 desires, and it is certain tha | | agadon ontallo ana tho rolovant |

The first ten subjects will be enrolled at the Coloplast Humlebæk Site DK001 (Sponsor). When these ten subjects have completed the first 7<sup>-1/+3</sup> days with the test product and completed the safety visit (V3) in proper compliance and with no unexpected events related to the test product, all following subjects can hereafter continue with enrolment and Test Period 2 at all sites.

The subjects, at other sites than DK001, will be invited for the Test Visit 1 during week 49-51 (December 2018) and for their Test Visit 2 during week 1 and 2 (January 2019), due to Christmas holiday, follow-up logistics and planning purpose. Hereafter, subjects will have 7-1/+3 days between their following visits.

The coordinating clinical manager will have close contact to each site during the recruitment period. The investigator at each site will notify the clinical manager of all planned inclusion visits and whenever a subject is enrolled. This will be done by mail and be site registration in a sheet for this purpose. When the coordinating clinical manager is aware that 25 subjects have been included, the recruitment will stop. Subjects who have been informed of the investigation and are reflecting on their participation may be included within the first 24 hours hereafter.

Enrolment period will be between 12-39 days for Test Period 1 and 28<sup>-4/+12</sup> days for Test Period 2. Site should however ensure that the visit windows are adjusted for the subjects to be terminated at last LSLV, at the latest.

#### 6.3.4. Subject withdrawal criteria

The subject is allowed to withdraw from the investigation at any time for whatever reason without any consequences for their future treatment outside the clinical investigation. Investigator may withdraw a subject from the investigation at any time if they judge it to be the subject's interest.

The investigator must withdraw a subject from the investigation due to:

- Non compliance with the CIP impacting the scientific integrity of the investigation
- If subject's safety and wellbeing is compromised by further participation.

Withdrawn subjects will not be replaced by new subjects.

A subject who is withdrawn from the investigation, for any reason, will be encouraged to contact the investigator if problems arise that the subject believes are related to the clinical investigation. Subjects who have not experienced any adverse events will not be followed up. For subjects who experience adverse events, see section 14.

#### 6.3.5. Point of enrolment

A subject is considered enrolled in the investigation when the written informed consent is obtained. The expected duration for each subject is described in section 6.1.

#### 6.3.6. Total expected duration of the clinical investigation

The dates below are approximate and no subjects will be enrolled before all required approvals have been obtained. Changes greater than ± 3 months will be notified to EC and regulatory authorities.

| Activity | Estimated time |
|-------------------------------|-----------------------------------|
| First subject enrolled | November 2018 |
| Last subject enrolled | December 2018 |
| Last subject completed (LSLV) | February, 12 <sup>th</sup> , 2019 |
| Final Report | February 2020 |

#### 6.3.7. Total number of subjects

Based on sample size calculations (see section 7.2) 21 one-piece users should be included in this investigation. However, to take potential drop-out into account a total of 25 one-piece users will be included (allocated a subject number).

#### 6.4. Procedures

#### 6.4.1. Clinical investigation-related procedures

See section 6.4.4 Flow-chart for a more detailed overview of the clinical investigation-related procedures at visit and 6.4.5 for a more detailed overview

#### Site visits

Before initiation of the clinical investigation, sponsor must be provided with key personnel's signed and dated curriculum vitae (not more than two years old) to verify their qualifications. Key site personnel are those, who conduct the clinical investigation and obtain subject data. Also, the sponsor will ensure that all site personnel are trained in the investigation procedures, how to complete the CRFs, procedure for reporting an adverse event and serious adverse event (how, when, to whom), and who to contact in case of emergency related to the investigational device.

#### Visit 0 (Information and Inclusion visit)

If a potential subject is interested in participating after the first contact, a visit (visit 0) will be arranged in a room reserved to ensure privacy and quiet surroundings at the investigators clinic/department. When arranging the visit, it will be ensured, that the subject has received the Subject Information Form prior to the visit. The subjects will receive both written and verbal information to ensure that the subject understand what was read and explained and can freely agree to participate in the investigation. The subject will, beforehand, also be informed about the possibility of bringing a companion to the informational visit and to any possible subsequent visits. During the visit the Investigator or delegated personnel will provide oral information about the investigation based on the Subject Information Form. The subjects have the right to wait 24h before deciding on participation. The information visit and the Visit 0 can be the same day.

If/when subjects decide to participate they will be asked to sign the Informed Consent Signature Form and other relevant forms (see section 13). If a subject so desires, and it is certain that it is understood what the investigation entails and the relevant forms have been signed the subjects are considered enrolled in the investigation. Enrolled subjects that fulfils the in- and exclusion criteria are allocated a subject number, and hereafter demographics, baseline data and concomitant medications is recorded by Investigator or delegated personnel.

Visit 0 and visit 1 can be combined.

#### Test visits (V1, V2, V4, V5 and V6)

During test visit 1, the subject will be introduced to the clinical app on how to complete the questionnaires and take pictures. At visit 2 the test products will be handed out. At this visit the subjects will be trained according to the IFU, in preparation of the product (e.g. hole size), preparation of skin before application (e.g. cleaning and wiping), application of product (e.g. correct position and applying pressure to the baseplate), removal of product and storage of the product.

At each test visit objective skin measurement will be done, the product changed at the visit will be collected for further analysis, pictures of cut product will be taken, stoma condition, skin condition and safety endpoints will be registered. At test visit 2 and 6 questions regarding feeling of security, handling, leakage scale and quality of life will be completed by subject. An output sample will be collected for further analysis at test visit 1 and 2. The output samples and products changed at the visit will be stored in a separately CP300 allocated freezer at site, and send on an ongoing basis to Coloplast A/S, Humlebæk, Denmark. The samples of output will not be stored longer than it takes to collect and analyse the samples. The sample will be destroyed directly after analysis.

At test visit 6 questions about product preference will be completed by subject.

#### **Product change**

At every product change the subjects will record reason for change, pain/discomfort, skin condition and use of accessories. Wear time of the product will be calculated from the time for product change registered in the app.

At every product change the subject will be asked to take a picture of the back side of the changed products (leakage), the peristomal skin and the cut product to be applied.

Subjects will also be informed about the possibility to contact a Coloplast nurse during the investigation, to ensure questions and experiences addressed answered properly. This will be a secondary contact person in addition to the study nurse at site.

#### Safety follow-up

To follow safety closely during the investigation, a safety visit (V3) is planned after one week of wearing the test product. The safety visit will, when logistically possible, be conducted by Sponsor at site, supported by Investigator or study nurse. The subjects will be asked about all experiences with their stoma during the investigation and other safety endpoints, following the safety interview guide (see Appendix 4). In addition, the product changed at the visit will be collected for further analysis.

To follow safety further, Sponsor might also wish to be presented at subjects' test visits. Sponsor will observe during the test visit and might ask the subject questions about experiences with their stoma during the investigation and other safety endpoints, following the safety interview guide (section 20.4).

#### Interview

The subjects will be offered to participate in two interviews. The interviews will be about the subjects experience with the test product and might include a change of product. The subjects can participate in the investigation without being interviewed. The interviews, or relevant parts, might be video recorded, tape recorded or photos might be taken. The subjects will be asked for consent, but can participate in interviews without completing video, tape or photos.

- Interview 1: at test visit 6 (at site) or within 14 days after termination (at home). If the interview is part of the test visit, Sponsor will be present during the test visit. At first, they will ask the subject unprobed questions to get their immediate response to the product. Hereafter, the subject can continue the test visit as usual. At the end of the visit, the interviewer will interview the subject following the interview-guide. If the subject has consented to photo, video and/or tape recording the interviewer might do so during relevant parts of the interview and test visit.
- **Interview 2**: a follow-up visit at home within three months after last patient out.

The information needed from interviews are estimated to be covered by up to 6-10 subjects, but all will be asked if they would like to participate, if more than ten are needed. If fewer than six subjects agree to be interviewed, we will settle for the number that have agreed. This has been decided since the main endpoints are covered in the CRF. It is known from experience that it is not always possible to perform all the interviews face-to-face due to logistics. In order, not to lose important information about the tested products, interviews may be by telephone / video call, in cases the interviewers cannot be present at the visits.

In addition, the study nurses and/or investigator may be interviewed during and/or within three months after termination of the investigation.

All interviews will be performed by Sponsor following an interview guide (Appendix 5).

#### Follow-up after the investigation

Subjects who do not have an ongoing AE, or are not participating in the second interview are not followed up on after termination of the investigation. For ongoing AEs at investigation termination, please see section 14.4. All subjects are encouraged to contact the Investigator or the associated Coloplast nurse after termination of

the investigation, if they experience problems that they believe are related to their participation. This is to ensure that any device-related events are documented and to safeguard the subjects' health.

#### 6.4.2. Activities performed by sponsor representatives

Sponsor or representative hereof (CRA/Monitor) will make a selection visit, site monitoring visits and site close out visit. At the selection visit Sponsor or representative hereof will ensure that the Investigator is qualified to conduct the investigation, is keen to participate, and has the time, resources and location to run the investigation. When the site has been selected to participate in the investigation, the Sponsor or representative will be responsible for:

- Training of investigator and delegated personnel in the investigation procedures, how to complete the CRF and how to report possible safety issues to Sponsor. All training will be documented by site and sponsor signing the Training Log. However, with any change of staff at site after the initiation, Principle Investigator is responsible for the training of the new staff.
- Identify and contact possible investigation subjects from Coloplast A/S's ostomy user database in Denmark and Sweden by letter, email or advertisement
- Support during the recruitment process
- Support during the test periods
- Monitor site as described in section 6.5 and the Monitoring Plan
- · Perform the interviews
- Collect and analyse data
- Equipment for measurements
- Comparator, test products, stoma scissors etc.
- Other equipment used during the visits (gloves, napkins, alcohol-gels etc.)

#### 6.4.3. Foreseeable factors that may compromise the outcome / results

Use of ostomy accessories may influence the actual performance of the test products. It is not known if accessories will have a "positive" or "negative" influence on the product performance. Subjects are asked not to use adhesive remover during the investigation as adhesive remover residues on the skin can interfere with the objective skin measurements such as TEWL. In addition, subjects who usually use a ring/seal will also be asked not to use these accessories during the investigation. This is to be able to understand the performance of the test products. However, for ethical reasons it is allowed that subjects that experience problems with removing the test products or leakage can use adhesive remover and rings/seals, respectively.

Some subjects enter the study using other accessories to minimise leakage under the baseplate. When this is part of the subject's standard care procedure these subjects may continue to use the accessories, they used when entering the study if they use the same accessories throughout the entire study period. It is important that a subject uses the same kind of accessories when testing the products as this gives the best conditions for comparing the performance of the products.

# 6.4.4. Flow-chart

Table 4: Chart showing the connection between visits and assessments

| Endpoint | Source | Performed<br>by | Inclusion<br>visit<br>(V0) | Visit 1<br>Test<br>visit<br>(V1) | Visit 2<br>Test visit<br>(V2) | Visit 3<br>Follow-<br>up/Safety<br>(V3) | Visit 4<br>Test<br>visit<br>(V4) | Visit 5<br>Test<br>visit<br>(V5) | Visit 6<br>Test<br>visit<br>(V6) | Follow-<br>up visit |
|---|---|---|---|---|---|---|---|---|---|---|
| Oral information | | Investigator <sup>1</sup> | X | | | | | | | |
| Written informed consent | Informed Consent Form | Subject | X | | | | | | | |
| Letter of Authority | Letter of Authority | Subject | X | | | | | | | |
| Consent to interview, including photo/video/tape record and three month contact | Informed Consent Form - Interview | Subject | X | | | | | | | |
| Declaration of Contraception | Declaration of contra-<br>ception Form | Subject | X | | | | | | | |
| Check of inclusion and exclusion criteria | Investigator Binder | Investigator1 | X | | | | | | | |
| Subject number allocated | | Investigator | X | | | | | | | |
| Registration of Baseline data | Investigator Binder | Investigator1 | X | | | | | | | |
| Assessment of subject wellbeing and compliance with CIP | NA | Investigator <sup>1</sup> | Х | Х | Х | Х | Х | Х | Х | Х |
| Collect used products changed at visit | Investigator binder √ | Investigatior1 | | Х | Х | X | Х | X | X | |
| Collect output sample | Investigator binder √ | Investigatior1 | | Х | Х | | | | | |
| Arrange dates for the next test visit | NA | Investigatior1 | X | X | Х | Х | X | Χ | | |
| Inform Clinical Manager about sched | | | | | | | | | | |
| | Investigator Binder | Investigatior <sup>1</sup> | | X | | | | | | |
| Comparator product hand-out | Device Accountability<br>Form | Investigatior <sup>1</sup> | | X | | | | | | |
| Subjects trained in how to prepare skin for the comparator product, and how to use, handle, cut and store the product, according to IFU. | Investigator Binder | Investigatior <sup>1</sup> | | Х | | | | | | |
| Test product hand-out | Device Accountability<br>Form | Investigatior <sup>1</sup> | | | Х | (X) | (X) | (X) | | |
| Subjects training: how to prepare skin for the test product, and how to use, handle, cut and store the product, according to IFU. | Investigator Binder | Investigatior <sup>1</sup> | | | Х | | | | | |
| Hand-out remuneration and obtain signature | Gift card reciept | Investiga-<br>tior <sup>1</sup> /subject | | Х | Х | Х | Х | Х | Х | (X) |
| Skin assessments and measurements | | | | | | | | | | |

| Endpoint | Source | Performed<br>by | Inclusion<br>visit<br>(V0) | Visit 1<br>Test<br>visit<br>(V1) | Visit 2<br>Test visit<br>(V2) | Visit 3<br>Follow-<br>up/Safety<br>(V3) | Visit 4<br>Test<br>visit<br>(V4) | Visit 5<br>Test<br>visit<br>(V5) | Visit 6<br>Test<br>visit<br>(V6) | Follow-<br>up visit |
|---|---|---|---|---|---|---|---|---|---|---|
| OBS!!! For TEWL, hydration and erythema: ea | | | e times in eac | A RESIDENCE OF THE PROPERTY OF THE PERSON OF | | | | | | |
| Acclimatisation 30 minutes | Investigator binder √ | Investigatior <sup>1</sup> | | X | X | | Х | Х | X | |
| Picture of peristomal skin | Investigator binder √ | Investigatior <sup>1</sup> | | Х | X | | Х | X | X | |
| (Light box + normal picture) | SD card | | | | | | | | | |
| Picture of reference spot | Investigator binder √ | Investigatior <sup>1</sup> | | X | X | | X | X | X | |
| (Light box + normal picture) | SD card | 200 | | | | | | | | |
| Picture of the cut product | Investigator binder √ | Investigatior <sup>1</sup> | | X | X | X | X | X | | |
| FIG. | SD card | 20 | | | | | | | | |
| TEWL | Investigator Binder | Investigator <sup>1</sup> | | X | X | | Х | X | X | |
| Inner circle (Four spots) | 17062 | 5840 | | | | | | | | |
| TEWL | Investigator Binder | Investigator <sup>1</sup> | | X | X | | Х | Х | Х | |
| Outer circle (Four spots) | 1000 | 557. | | | | | | | | |
| TEWL | Investigator Binder | Investigator1 | | X | Х | | X | Χ | Х | |
| Reference spot | 1771 | 1744 | | | | | | ., | | |
| Hydration | Investigator Binder | Investigator <sup>1</sup> | | X | X | | X | Χ | X | |
| Inner circle (Four spots) | 5255 | 10793 | | | | | | | | |
| Hydration | Investigator Binder | Investigator <sup>1</sup> | | Х | X | | Х | Х | Х | |
| Outer circle (Four spots) | | - | | | | | | | | |
| Hydration | Investigator Binder | Investigator1 | | Х | X | | Х | Х | Х | |
| Reference spot | STOREST AND SERVICES AND SERVIC | Production for the area with | | 242,340 | 3500,000 | | 5000 | 100000 | \$95,859 | |
| Erythema | Investigator Binder | Investigator1 | | Х | X | | Х | Х | Х | |
| Inner circle (Four spots) | | responsible to bride to be supported | | 25500 | 1000000 | | 500 | 1500,000 | \$95385) | |
| Erythema | Investigator Binder | Investigator1 | | Х | Х | | Х | X | Х | |
| Outer circle (Four spots) | | PRICE CONTRACTOR OF THE PRICE O | | 0.9652 | 8-980 | | 25576 | 31,080 | 275927 | |
| Erythema | Investigator Binder | Investigator1 | | Х | Х | | Х | Х | Х | |
| Reference spot | | and second to Sussessi | | 5.759365 | 5-62565 | | 935 | 2-030/0 | NAMES | |
| Endpoints completed by subject at visits | | | Service Servic | | - | - | | ä. | | |
| Feeling of security, handling, quality of life, leak- | Subject questionnaire | Subject | | | Х | | | ** | Х | |
| age scale questionnaire | | • | | | | | | | 7.00.00 | |
| Skin condition – skin complications | Subject questionnaire | Subject | | Х | Х | | | | Х | |
| Skin condition – change of skin complications | Subject questionnaire | Subject | | | Х | | | | Х | |
| Stoma condition - questions | Subject questionnaire | Subject | | | Х | Х | Х | Х | Х | |
| Preference | Subject questionnaire | Subject | | | | | | y zeven | X | |
| Endpoint | Source | Performed<br>by | Inclusion<br>visit<br>(V0) | Visit 1<br>Test<br>visit<br>(V1) | Visit 2<br>Test visit<br>(V2) | Visit 3<br>Follow-<br>up/Safety<br>(V3) | Visit 4<br>Test<br>visit<br>(V4) | Visit 5<br>Test<br>visit<br>(V5) | Visit 6<br>Test<br>visit<br>(V6) | Follow-<br>up visit |
|---|---|---|---|---|---|---|---|---|---|---|
| Endpoints registered by Investigator <sup>1</sup> | | | | | | | | | | |
| Adverse events incl. supplementary information | Investigator Binder | Investigator1 | | X | Х | X | Х | Х | Х | |
| Device Deficiencies | Investigator Binder | Investigator1 | | X | X | X | Х | Χ | X | |
| Concomitant medication | Investigator Binder | Investigator1 | Х | X | Х | X | X | X | X | |
| Skin condition – Discoloration/Damage/Raised tissue | Investigator Binder | Investigator <sup>1</sup> | | Х | Х | | Х | Х | Х | |
| Skin condition - Change in skin complications | Investigator Binder | Investigator <sup>1</sup> | | | Х | | | | Х | |
| Qualitative data | | Table State of the | | | A | | | | No. | |
| Safety interview | Interview notes | Sponsor <sup>1</sup> | | | | Х | | | | |
| Interview (termination) | Interview notes <sup>2</sup> | Sponsor <sup>1</sup> | | | | | | | Х | |
| Interview (follow-up) | Interview notes <sup>2</sup> | Sponsor <sup>1</sup> | | | | | | | | Х |

<sup>&</sup>lt;sup>1</sup> Qualified site personnel can perform investigation related tasks as investigator representatives. This delegation will be documented in the "Site Personal Signature and Delegation List" for each site. All investigators and investigator representatives will receive oral and written training in all investigation related tasks before they can begin any investigation related tasks. The training will be documented in the Clinical Investigation Training Log.

<sup>2</sup>The interview notes will be stored at the secure Coloplast User Insight Drive.



#### 6.4.6. Randomisation Procedure

Not applicable since no randomisation will take place

## 6.4.7. Blinding

The investigation is not blinded because the test product and SenSura® Mio are visible different from each other. If the subjects have a preconceived attitude to the test products or SenSura® Mio bias could occur for all subjective parameters.

## 6.4.8. Case Report Forms

The CRFs are printed and supplied by Sponsor. The CRFs are printed on NCR paper in order to have one copy for investigator and one copy for sponsor (original copy). A CRF is provided for each subject. It is the responsibility of the Investigator that all data are entered promptly and correctly.

Each CRF have printed instructions for completion.

The CRF will be filled in by the subject and by the investigator/relevant staff, who have signed the Site Personnel Signature and Delegation List and Clinical Investigation Training Log. It will be the responsibility of investigator that all measurements and observations are correctly noted with a pen (permanent writing utensil) in the CRF.

The Case Report Forms for each subject will be divided in three parts:

- **Investigator Binder;** Investigators registration of inclusion and exclusion criteria, baseline data, skin measurements, stoma condition, skin condition and safety endpoints at visits.
- **Subject questionnaire**; Subjects registration of feeling of security, handling, quality of life, leakage scale questionnaire and preference at visits.
- Subject diary and paper); Subjects completion of reason for change, skin condition, use of accessories, pain/discomfort, and subject pictures will be registered

Qualitative endpoints (interviews) will be registered as notes, and will not be part of the CRF. Other endpoints than the above mentioned will be registered directly from source to the data base.

Any correction in the CRF must be clearly signed and dated by authorised site personnel. The entry corrected must be crossed out so that the entry is still legible.

#### Example 1: Example 2:



Figure 4 Two examples of how to make corrections in the CRF

The investigator will keep a separate list with the subject ID numbers, names and addresses in a locked room. Only data referred to in this clinical investigation plan will be recorded in the CRFs.

CRFs will be collected and send to site continuously by Monitor after completed monitoring and sign of by Investigator.

#### 6.4.9. Concomitant treatment

Concomitant treatment, including medication, will be registered in the CRF.

Subjects are not allowed to use ring/seals, unless they can't do without. See also section 6.4.3 for foreseeable factors.

## 6.5. Supplementary material and equipment

The Sponsor will provide the sites with supplementary materials for this investigation. Supplementary materials would be:

- CRFs
- \_
- Skin measurements equipment
- Camera with lightbox
- Camera
- Subject toilet bags including stoma guide, scissor, pen, disposal bags etc.
- Nurse kits including disposal bags, gloves, gauze, disinfection gel etc.

#### 6.6. Monitoring Plan

Coloplast representatives will review data centrally to identify potential issues to determine a schedule of onsite visits for targeted review of study records.

For safety reason the Coordinating Investigator, a delegate hereof or equivalent competent Coloplast representatives will monitor the subjects' stoma if relevant by visiting the sites when subject visits are performed.

Coloplast representatives must be allowed to visit all study site locations periodically to assess the data quality and study integrity. On site, they will review Study CRFs and directly compare them with possible source documents, discuss the conduct of the study with the investigator, and verify protocol compliance, and that the facilities remain acceptable. CRF pages and/or subject files at site may serve as the source documents.

Signed ICF, Subjects identity any AE/SAE and Concomitant Medication will be monitored 100 %. All entered data in the CRF will be reviewed for completeness and for relevant purpose.

When a site has been visited for monitoring a monitoring report is written to document the status of the study at site and to ensure the rights, safety and well-being of the subject are protected, and that all data obtained by the site is consistent with the protocol.

Detail for the monitoring visits are described in the Monitoring Plan. The Monitoring Plan explain the type of visit relevant for the study and why they are performed, the frequency of the monitoring visits, and the timeline for the Reports.

The study may undergo audit and/or inspection, which allow access to CRFs, source documents, other study files, and study facilities. The audit/inspection will be announced when relevant. Audit reports will be kept confidential.

The investigator must notify Coloplast promptly of any inspections of the study scheduled by regulatory authorities, and forward copies of inspection reports to Coloplast.

#### 6.6.1. Source data verification

The Monitor will ensure proper access to all Source Data due to local regulations.

A Source Data Specification Form, detailing the location of all source data (Paper CRF, Subject diary Interviews incl. video/tape recordings and photos (if applicable)) for each data point, shall be completed at the initiation visit for the investigational site to document what is source data for the data collected at each site. This Source Data Specification Form must be signed and dated by the Investigator and the Monitor to verify the agreement between the two parties and when this Source Data Specification Form was agreed. Source data verification must be performed, -per monitoring plan for all 25 expected enrolled subjects.

For all subjects, the following will be 100% source document verified:

- Informed Consent Forms
- Inclusion and exclusion criteria
- Letter of Authority Form
- Declaration of Contraception Form
- Inclusion number /
- Primary and explorative endpoints
- All protocol-defined adverse events (AE), ADE, SAE, SADE

Furthermore, the following will be reviewed/monitored for completeness and consistency:

- All Data entered in the CRF
- Deviations
- Subject diary
- Device Accountability

At the discretion of the monitor and in consultation with the Clinical Manager additional data may be reviewed in case of quality concerns such as:

- Non-compliance and data quality issues
- Number of and/or type of unreported adverse events observed during source data verification
- Number of and/or type of deviations
- Number of unresolved queries/data clarification forms

At the completion of the monitoring visit, the monitor will meet with the investigation coordinator and/or Principal Investigator, if necessary, to review and discuss the monitoring findings. In addition, the monitoring accomplishments and findings will be reviewed by the Coloplast study team and Clinical manager or designee to assess corrective action measures as needed.

The Informed Consent forms – and the Letter of Authority form - and compliance with the inclusion and exclusion criteria, as well as all AEs, are verified 100% for completion at the correct time. All CRFs are monitored for incomplete data and incorrect data. Furthermore, all events that occur during the investigation period are registered in the CRF and followed up by the Investigator.

Only the Investigator, delegated site personnel and representatives of the sponsor will have access to all CRFs. The subjects will have access to their own CRF (however, see also section 12.3).

Representatives of the sponsor are: Data manager, Coordinating Clinical Manager, Clinical Managers, Scientific Manager and the medical adviser. In relevant situations, the data responsible can allow others to access the CRFs.

# 6.6.2. Other methods for data quality assurance

The sponsor, sponsor's representative and/or investigational sites may be inspected by competent authorities or their representatives and likewise may be audited per Coloplast's internal quality audit plan and procedures. The investigator allows access to source data, medical records and other relevant documents for this study both for monitoring, audit and/or inspections from the Ethics Committee and authorities from other countries.

#### 7. Statistical considerations

# 7.1. Statistical design, method and analytical procedures

Definition of analysis populations:

The ITT population (full analysis set) will be constituted by all included subjects who:

- · Have provided valid informed consent
- Have valid information for at least one of the endpoints

Invalid individual data points may be omitted from analysis even though the corresponding subject is part of the ITT population. Any exclusion of data points will be documented.

The Safety population (basis for presentation of AEs) will constitute by subjects who have given informed consent.

A formal PP population is not planned due to the explorative nature of the investigation. Considering the data obtained it might however be considered to make additional explorative analyses based on a subset of the ITT population.

#### Analysis of the primary endpoint

The primary endpoint is TEWL measured at 4 spots (up, down, left and right) around the stoma in the inner circle at steady state. For each subject 3 repeated measurements will be made for each spot and at each test visits at site for products worn in the 2 test periods. The comparison in TEWL between the 2 products is used to evaluate the primary objective of the investigation.

A linear mixed model will be applied to the log transformed TEWL data. The model will include a fixed effect of product (comparator and test product). Further the model will include:

- a random effect of subject
- · a random interaction effect of product and subject
- · a random interaction effect of spot in the inner circle and subject
- a random interaction effect of product, spot and subject
- · a random interaction effect of product, visit and subject
- a random interaction effect of product, spot, visit and subject.

If the assumption of steady state for the test product is not reached after 2 weeks, the analysis can be performed with only test product data from visit 5 and 6 (3 and 4 weeks).

From this model the difference in TEWL between products will be estimated. As TEWL is analysed log transformed the estimated differences on log-scale will be back-transformed to the original scale as estimated ratios.

#### Analysis of the exploratory endpoint

To include the information from the reference spot on the abdominal site, all the above described analyses will be performed as explorative analyses with the dependent variable as the difference between the endpoint and the mean of the corresponding measurements from the reference spot.



From this model the difference in leakage area and distance between products will be estimated

As this is the first time the "skin condition endpoints (Assessed at every product change)" have been included in a study, the data will be used to evaluate how the results can be summarised, interpreted and analysed in upcoming studies.

As it is an exploratory study no adjustment for multiple testing will be applied.

Photos will be evaluated visually in this exploratory study. Collected baseplates and output samples will not be evaluated statistically.

All other endpoints will be listed or summarized by descriptive statistics. Additional summaries can be made for endpoint only collected in the steady state periods.

## Analysis of safety endpoints

Adverse events will be listed. Results from the safety questions (Safety questions about changes in stoma normalities and additional pain questions) will be listed and/or summarized by descriptive statistics.

All statistical analyses will be made with SAS version 9.4 (SAS Institute Inc., Cary, NC).

#### 7.2. Sample size

The primary endpoint is TEWL measured at four spots in the inner circle (up, down, left and right) around the stoma. For each subject three repeated measurements will be made for each spot at two different days for products worn in test period 1 and for three different days for test period 2.

Part of the primary objective is to compare TEWL measured at the inner circle around the stoma when subjects are exposed to own output using comparator product and using the test product. The comparison will be performed by a model using all available TEWL data from the inner circle.



- a random interaction effect of spot in the
- a random interaction effect of product, s
- · a random interaction effect of product, vi
- a random interaction effect of product, s
- and the residual accounts for

In Table 5 the needed sample size is calculated by simulation for varying values of the true ratio in TEWL and for different values of the power to demonstrate that the ratio is significantly different from 1 (that the 95% confidence interval excludes 1).

Table 5: Subjects needed for comparing mean TEWL for two products



Based on the numbers in the table, 21 subjects should test ratio between the comparator product and a test product is take a potential drop-out into account it is recommended to include a total of 25 1-pc subjects.

# 7.3. Level of significance and power

Statistical tests will be carried out as two sided tests on a 5% level of significance. For information regarding the power, see the above section.

#### 7.4. Drop-out

The sample size has been calculated based on an assumed drop-out rate of 20%. Due to the exploratory nature of the study, drop-out subjects will not be replaced.

#### 7.5. Pass/fail criteria

No formal success criteria are applied in this explorative investigation. The investigation will provide valuable insight into how the peristomal skin reacts

# 7.6. Interim analysis

No interim analysis is planned for this study.

# 7.7. Statistical reason for termination of investigation

There is no reason to terminate the investigation based on statistical considerations.

## 7.8. Deviation(s) from statistical plan

Any deviations from the statistical plan will be documented in the clinical report.

# 8. Data management

## 8.1. Data review, database cleaning, and issuing and resolving data queries

Data management and statistical analyses is carried out by Medical Affairs, Coloplast A/S.

To ensure correct data entry, data is entered twice (double data entry). Data management is responsible for control of data consistency and also for completeness of data from each subject.

Discrepancies are listed in Data Query Forms (DQF), and the Investigator is responsible for solving these promptly. When all DQFs are solved the database is locked and the final statistical analyses are performed.

# 8.2. Verification, validation and securing of electronic clinical data systems

EXPeRT Data Management, version 5.0.05 system delivered by OmniComm Systems Inc. is used for data management. The system is designed to be compliant with the requirements of 21 CFR part 11. It is a validated data management system allowing only qualified and trained personnel to enter the system.

For collection of the subject diary data, Coloplast A/S uses a newly developed clinical trial application developed by "Blue Fragment".

# 8.3. Data retention

The sponsor file must be archived for a minimum period of 5 years after the final clinical investigation report has been signed.

All investigation site documents must be archived for a minimum period of 5 years after the final clinical investigation report has been signed. The monitor is responsible for informing the investigator and the CTM if this period should be longer for their sites according to local regulation.

# 9. Amendments to the CIP

Any significant changes to the CIP are:

- Agreed between sponsor, PI(s) and the coordinating investigator.
- Justified in a statement included in the amended section and the version number and date of amendment must be documented.
- Registered in the Change Log.
- Notified to or approved by the EC before implementation
- Notified to or approved by the regulatory authorities before implementation

Example of significant change: Changes of inclusion criteria, endpoints or assessment methods.

# 10. Clinical Investigation Plan deviations

#### 10.1. Deviations

Deviations to Clinical Investigation Plan occurs when the activities during the clinical investigation diverge from the Ethic committee approved investigation plan.

A deviation does not increase risk or decrease benefit or; does not have a significant effect on the subject's rights, safety or welfare; and/or on the integrity of the data.

Examples of deviations:

- Vital signs obtained prior to informed consent
- Partly completing required tests

The Investigator is not allowed to deviate from the Clinical Investigation Plan unless under emergency circumstances and to protect the rights, safety and well-being of the subject(s).

Deviations must be reported to sponsor and deviations affecting the scientific aspect of the investigation or the safety of the subject are reported to the Ethical Committee by sponsor.

If any deviations and/or violations to the investigation plan are detected, the Clinical Manager will complete a Deviation/Violation Form and inform/discuss with the Principal Investigator immediately.

#### 10.2. Violations

Violations to the Clinical Investigation Plan occurs when there is divergence from the Ethical Committee approved investigation plan (a deviation) that also:

- · Reduces the quality or completeness of the data
- · Impacts a subject's safety, rights or wellbeing
- · Affects the scientific integrity

#### Examples of violations:

- Inadequate informed consent
- Enrolment of subjects not meeting the inclusion / exclusion criteria
- · Initiation of study procedure prior to completion of informed consent
- Unreported SAE's
- Repeated deviations of the same nature
- Falsification

If any deviations and/or violations to the investigation plan are detected, the Clinical Manager will complete a Deviation/Violation Form and inform/discuss with the Principal Investigator immediately.

In case of continued or repeated violations affecting the scientific aspect of the investigation or the subjects' rights, safety and well-being sponsor will disqualify the PI from further participation in the investigation.

The Clinical Manager must report all violations detected during a monitoring visit in the Periodic Monitoring Report.

# 11. Device Accountability

All access to the investigational devices used in the clinical investigation is controlled by storage procedures and device accountability logs as described below. The investigational devices must only be used in this clinical investigation and only according to the Clinical Investigation Plan.

Sponsor keeps a device accountability log that states the physical location of all investigational devices from shipment of investigations devices to the investigational sites until return of or disposal.

The Investigator or a delegate hereof keeps records documenting the receipt, use and return and disposal of the investigational devices, which includes:

- Date of receipt.
- Identification of each investigational device (batch no./serial no./uniqe code).
- The expire date, if applicable.
- Subject identification.
- The date on which the investigational device was distributed to the subject.
- The date on which the investigational device was returned/explanted from the subject
- The date of return unused, expired or malfunctioning investigational devices

# 12. Statement of compliance

The clinical investigation is conducted in accordance to:

- Ethical principles that have their origin in the Declaration of Helsinki, 1964, Last amended at the 59th WMA General Assembly, Seoul, October 2008.
- MDD 93/42/EEC as amended by Directive 2007/47/EC (commonly known as the Medical Device Directive).
- ISO 14155:2011 "Clinical Investigation of medical devices for human subjects Good clinical practices".
- Any applicable regional or national regulations

# 12.1. Ethics committee and regulatory authorities

The CIP and/or other relevant documents are submitted to the appropriate EC(s) and regulatory authorities. This clinical investigation will not begin until the required approval from the EC and regulatory authorities have been obtained. Any amendment to the protocol will be submitted to the same EC(s) and regulatory authority. Sponsor will notify the relevant regulatory authority and EC(s) concerned of the end of the clinical investigation. Approval from the Danish Protection Agency is not necessary as this clinical investigation is done by a private company and therefore is exempted from notification.

## 12.2. Data protection

All information collected during this investigation is owned by Coloplast and is kept strictly confidential. Subjects are identified by an investigation number and the investigation monitor has access to subjects' notes/documentation for source data verification. Monitoring and monitoring findings will be documented in a report to explain and document that the rights and well-being of the subjects are protected, that the reported data are accurate, complete and verifiable from source documents, and that the conduct of the investigation is following the currently approved Clinical Investigation Plan (CIP), including amendments, and with the applicable regulatory requirements. The reports have no subject identification and are kept confidential during the conduct of the investigation and during archiving for 6 years. Subjects remain anonym for data analysis, as the data is blinded correspondingly in the data analysis.

Should the investigation require future review, relevant ethics committees and Coloplast Internal Audit performer will be allowed access to all relevant information for audit purposes.



Coloplast complies with applicable data privacy law, including the <u>EU General Data Protection Regulation</u> ("GDPR"). Under GDPR the legal basis for Coloplast's collection and use of the personal information is for the purpose of analyzing samples, and all data collected in this clinical investigation to innovate and improve Coloplast's stoma products.

Coloplast protects all personal information and will only allow it to be used for the mentioned purposes related to only this clinical investigation.

Each subject is entitled to get access to all the data and to have rectified any inaccurate data Coloplast is processing about the subject. All data are collected based on the consent each subject has given when being eligible and enrolled in the investigation. The subject is entitled to withdraw any such consent at any time, and

Coloplast will then cease to use such personal information for further innovation and improvement of stoma products. The already data collected and handled in the investigation will not be retired.

For further information please see Coloplast's Global Privacy Notice (<a href="www.coloplast.com/global/privacy-no-tice">www.coloplast.com/global/privacy-no-tice</a>).

# 12.3. Indemnity



#### 12.4. Financial conditions

The clinical investigation is initiated and sponsored by Coloplast A/S.

Coloplast A/S will pay all investigators involved in the clinical investigation for their time and resources spent on site to comply with the Clinical Investigation Plan. All financial agreements with the investigation sites involved in the clinical investigation will be specified in a sponsor investigator agreement. All investigator participating in this clinical investigation are employed at private clinics conduct clinical investigations.



# 13. Informed consent process

Written informed consent is obtained at visit 0 (inclusion visit) from all subjects participating in the investigation after thorough written and verbal information. The informed consent process takes place in a room reserved for ensuring privacy and quiet surroundings at the investigator's department. The subjects will receive both written and verbal information about the possibility of bringing a companion to the visit and to any possible subsequent visits.

The information is given by the investigator or a delegate hereof in the subjects' native non-technical language. Each subject will be fully informed about the aim of the investigation, procedures, potential risks or inconveniences and/or expected benefits and have a minimum of before deciding on participation. The subjects will be

informed that their participation is voluntary and that they may leave the investigation at any time, without this having any influence on their further treatment.

If the subject decides to participate in the clinical investigation, the subjects will be asked to sign a Consent Form, in which the subject consent to participate under the circumstances described in Subject Information Form.

When signing, the Consent Form the subject accept to pass all data and information, received from the subject by the investigation physician or investigation staff during the investigation, to Coloplast A/S, and/or representative hereof, relevant competent authorities and to a third party including those in countries outside the European Union. The consent for access to the parts of the subjects medical records, that are relevant to the investigation, covers the investigation period and an additional five years. This is to verify that collected data are accurate, and that the investigation is being carried out as planned and in agreement with the current laws and regulations.

All parties involved in this clinical investigation, also including relevant authorities, are governed by confidentiality about the information, they might be aware of. All collected data and information will be kept and stored confidential and in an anonymous form by Coloplast A/S who is data responsible. The investigation physician will use an investigation subject ID number to identify the subject.

In addition, the subject will be asked to sign the following documents:

- Subjects must also sign a power of attorney, which permits the sponsor and the authorities to gain access to data registered as part of this investigation, including their medical records if necessary.
- Woman in the childbearing age, will be asked to sign a Declaration of Contraception Form, which confirms that the subject do not plan to get pregnant during the investigation period, and that the subject will use birth control during the investigation.
- In addition, the subject will be asked if they would like to participate in two interviews, as described elsewhere in this protocol. It is voluntarily to participate in interviews, and the subject can participate in the clinical investigation without being part of the interviews.
- If the subject consent to interviews, the subject will be asked to consent to have pictures taken, video or tape recorded during parts or during the whole interview. It will not be possible to identify the subject from the pictures, video and tape records taken, and the participation is voluntarily. The subject can participate in the two interviews without having any pictures, video or tape records taken.

The informed consent signature form and the above-mentioned form includes personally dated signatures of the subject and the Principle investigator or a delegate hereof responsible for conducting the informed consent process. A copy of all signed forms will be provided to the subject.

If new information is to be given during the investigation, sponsor will inform the investigators, and the new information is given to the subjects by the investigator. If new information becomes available that can significantly affect a subject's future health and medical care that information will be provided to the subject in written form. Clinical Manager is responsible for writing the information and providing it to investigators that will further provide it to the subjects. If applicable, all affected subjects shall be asked to confirm their continuing informed consent in writing.

This procedure also applies to informed consent obtained from a subject's legal representative. The procedure cannot waive the subjects' legal rights.

# Adverse Event Device / No No Adverse Event (AE) Is it serious? procedure related? Yes Yes Adverse Device Serious Adverse Effect (ADE) Event (SAE) Device / procedure related? Yes Serious Adverse Unanticipated No Anticipated? Device Effect SADE (SADE) Yes Anticipated SADE

# 14. Adverse events, serious adverse events and device deficiencies

Figure 5: Adverse event flow

#### 14.1. Adverse events

#### 14.1.1. Adverse event

An adverse event is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other parties, whether or not related to the medical device(s), or the procedures involved. This could include events such as headache or dizziness.

#### 14.1.2. Adverse device effect

An adverse event, which is related to the use of the investigational medical device, is an adverse device effect, and should be marked as related or possibly related on the adverse event form.

The definition of an adverse device effect includes any event resulting from insufficiencies or inadequacies in the instruction for use, malfunction of the device, use error or from intentional misuse of the device. Table 6 lists anticipated adverse device effects that may occur.

Table 6 Anticipated adverse device effects and their likely incidence rates

# ANTICIPATED ADE Peristomal skin irritation (incl. mechanical trauma) Allergic peristomal skin irritation (dermatitis) Irritated stoma (incl. strangulation of stoma)

The definition of an adverse device effect includes any event resulting from insufficiencies or inadequacies in the instruction for use, malfunction of the device, use error or from intentional misuse of the device.

Please see section 4.2 for an overview of anticipated risks.

Temporary redness upon removal of the baseplate is not considered to be an adverse device effect. However, an abnormal development in the intensity or duration of redness should be considered an adverse device effect. A development in redness after removal of the baseplate is considered abnormal, when the intensity of redness is not decreased after five-ten minutes after the baseplate has been removed.

# 14.2. Device deficiency

A device deficiency is the inadequacy of the investigational medical device with respect to its identity, quality, durability, reliability, safety or performance. This includes malfunctions, misuse or use errors and inadequate labelling.

Primary and explorative endpoints that are measured during this investigation will not be required to be reported as device deficiencies.

#### 14.3. Serious adverse events

#### 14.3.1. Serious adverse event

A serious adverse event is an adverse event that:

- · Led to death,
- Led to a serious deterioration in health of the subject that either resulted in:
  - 1) a life-threatening illness or injury, or
  - 2) a permanent impairment of a body structure or a body function, or
  - 3) required in-patient hospitalization or prolongation of existing hospitalization, or
  - 4) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
- Led to fetal distress, fetal death or a congenital abnormality or birth defect.

This includes device deficiencies that might have led to a serious adverse event if:

- · Suitable action had not been taken, or
- Intervention had not been made, or
- Circumstances had been less fortunate.

These are handled under the serious adverse event reporting.

Planned hospitalization for a pre-existing condition, or a procedure required by the CIP, without serious deterioration in health, is not considered a serious adverse event.

#### 14.3.2. Serious adverse device effect

A serious adverse device effect is an adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event.

# 14.3.3. Anticipated serious adverse device effect

Anticipated serious adverse device effect is any event that by its nature, incidence, severity or outcome has been previously identified in the risk analysis report.

## 14.3.4. Unanticipated serious adverse device effect

An unanticipated serious adverse device effect is a serious adverse device effect which by its nature, incidence, severity or outcome has not been identified in the current version of the risk analysis report.

## 14.4. Medical care of subjects

Principal investigator shall ensure that adequate medical care is provided to a subject experiencing an adverse event during and after participation in the clinical investigation. All serious adverse events will be followed until a resolution is addressed.

The current status of all ongoing adverse events is documented during site close-out.

## 14.5. Reporting and timelines

#### 14.5.1. Investigators reporting responsibilities

PI must assess all (S)AE's that occur at his/her site.

- All serious adverse events and serious adverse device effects must be reported to Sponsor immediately, but no later than three calendar days, after Investigator or other site personnel's awareness of the event.
   When reporting the SAE the relationship to the test product shall be described whether the event is considered:
  - Not related, the event has no temporal relationship with the use of the test product or the procedures.
  - Unlikely related, the relationship with the use of the test product seems not relevant and/or the
    event can be reasonably explained by another cause, but additional information may be obtained.
  - Possible related, the relationship with the use of the test product is weak but cannot be ruled out completely. Alternative causes are also possible (e.g. an underlying or concurrent illness/ clinical condition or/and an effect of another device, drug or treatment). Cases were relatedness cannot be assessed or no information has been obtained should also be classified as possible.
  - Probable related, the relationship with the use of the test product seems relevant and/or the event cannot reasonably be explained by another cause, but additional information may be obtained.
  - Causal relationship, the event has a temporal relationship with the test product use/application or procedures.
- A device deficiency that could have led to a serious adverse event but did not because suitable action was
  taken, intervention had been made or because of fortunate circumstances should be reported to Sponsor,
  immediately, but no later than three calendar days, after Investigator or other site personnel's awareness of
  the event.
- New findings and/or updates in relation to already reported serious events should also be reported to Sponsor within three working days.

• Device deficiencies and all adverse device effects must be reported to sponsor within 10 days.

All above events must be reported by use of the relevant adverse event/serious adverse event/device deficiency form.

All above events must be reported by use of the relevant adverse event/serious adverse event/device deficiency form.

Please report to:

Clinical-studies@coloplast.com



# 14.5.2. Sponsors reporting responsibilities

It is the responsibility of sponsor to ensure that the following are reported to national regulatory authorities immediately and ethics committee (if required), but no later than seven calendar days following the date of awareness by Sponsor.

- All serious adverse events.
- · All serious device effects.
- All device deficiencies that could have led to serious adverse events but did not because suitable action was taken, intervention had been made or because of fortunate circumstances.
- New findings and/or updates in relation to already reported events.

If the serious adverse event results in imminent risk of death, serious injury, or serious illness that requires prompt remedial action for other subjects, users or other persons or a new finding to such a serious adverse event, sponsor must immediately but no later than two calendar days after awareness by sponsor report the event to national regulatory authorities.

It is the responsibility of sponsor to inform all investigators in writing within ten working days if device deficiencies, adverse events, adverse device effects, near-incidents, serious adverse events, serious adverse device effects or unanticipated serious adverse device effects lead to corrective actions (e.g. change of IFU).

# 15. Suspension or premature termination of the clinical investigation

Sponsor may suspend or prematurely terminate an investigation site or the entire clinical investigation for documented significant reasons.

If a suspicion of an unacceptable risk to subjects develops during the clinical investigation, Sponsor will suspend the investigation while the risk is assessed. Sponsor will terminate the investigation if an unacceptable risk is confirmed. Sponsor will ensure that the premature termination will be justified in writing and will promptly inform the regulatory authorities and relevant EC(s). If monitoring or auditing of the clinical investigation identifies serious or repeated deviations at one of the participating investigation sites, sponsor will suspend or terminate the particular investigation site. The sponsor or investigator will inform the regulatory authority as appropriate and notify the EC about the termination of the site.

If suspension or termination of the clinical investigation occurs, the investigator(s) will promptly inform the enrolled subjects. Sponsor will provide resources to fulfil the obligations from the CIP for follow-up of the subjects as necessary.

# 16. Clinical investigation report

At completion of the investigation sponsor is responsible for writing the clinical investigation report. The report is retained on file. The report contains a critical evaluation of all data, which have been collected during the investigation. The report describes the methodology and design and a data analysis, including statistical preparation and conclusion.

Sponsor and national coordinating investigators must sign the final version of the clinical investigation report or an affidavit, indicating their agreement with the contents. If no coordinating investigators are appointed, then the signatures of the principal investigators should be obtained.

The clinical investigation report will be submitted to relevant Ethics Committees and regulatory authorities within one year after last subject out.

# 17. Publication policy

# 17.1. General

Coloplast, sponsor, is referring to the internal document 'Clinical Publication Policy' that will be available for internal and external persons involved in the publication process.

The investigation will be registered on a public accessible database, e.g. www.ClinicalTrial.gov, before recruitment of the first subject. The results of the investigation, positive as well as inconclusive and negative will be published in the same public accessible database. The subjects' identity will remain confidential. Publication of results in the database will be conducted per the law of personal data protection and will be initiated as soon as scientifically acceptable, however, within one year after the last subject has completed the investigation. Data from the investigation is considered confidential until it is published per the conditions of this CIP and the 'Clinical Publication Policy'. Sponsor may publish anonymous single subject case stories (or public, if the subject consents) at any time during and after the investigation. The identification of the participant must not be possible. Sponsor reserves the right to use the data (published and unpublished) for reimbursement or regulatory purposes.

# 18. Bibliography

[1] Coloplast-A/S, "Investigator's Brochure CP300")".

[2] M. H. S. M. P. R. A. Y. L. M. K. J. Janet Stoia Davis, "Factors impairing quality of life for people with an ostomy," *gastrointestinal Nursing*, 2011.

# 20. Appendix

# 20.1. Appendix 1: LOCAL CHANGE LOG

A Local Change Log should be created per country specific CIP (e.g. one Local Change Log for French CIP and one Local Change Log for Danish CIP).

| VERSION<br>NUMBER | ISSUED BY<br>(INITIALS) | COMMENTS (MAJOR CHANGES SINCE LAST REVISION) |
|---|---|---|

# 20.2. Appendix 2: Leakage scale questionnaire

# Emotional impact

When you thought about your ostomy device and the risk of leakage, what emotions did you feel?

| In the last 7 days, due to leakage or worry about leakage… | All of the time | Often | Sometimes | Rarely or never |
|---|---|---|---|---|
| I felt panic | 0 | 1 | 2 | 3 |
| I felt stressed out | 0 | 1 | 2 | 3 |
| I felt more afraid about leaks in the future | 0 | 1 | 2 | 3 |
| I felt worry | 0 | 1 | 2 | 3 |
| I felt frustrated | 0 | 1 | 2 | 3 |
| I felt embarrassed | 0 | 1 | 2 | 3 |
| I felt worried that I might leak | 0 | 1 | 2 | 3 |
| l couldn't sleep | 0 | 1 | 2 | 3 |
| I kept waking up at night to check my stoma | 0 | 1 | 2 | 3 |
| I kept checking my ostomy bag to see if I have leaked | 0 | 1 | 2 | 3 |

# Usual and Social activities

When you thought about your ostomy device and the risk of leakage, how did it affect your activities?

| In the last 7 days due to leakage or worry about leakage | All of the time | Often | Sometimes | Rarely or never | Not applicable |
|---|---|---|---|---|---|
| I decided to stay at home | 0 | 1 | 2 | 3 | 9 |
| I couldn't do light activities | 0 | 1 | 2 | 3 | 9 |

| I changed my plans | 0 | 1 | 2 | 3 | 9 |
|----------------------------------------------------------|---|---|---|---|---|
| I was unable to go out and meet family and friends | 0 | 1 | 2 | 3 | 9 |
| I avoided close physical contact with family and friends | 0 | 1 | 2 | 3 | 9 |
| I did not want to see people | 0 | 1 | 2 | 3 | 9 |
| I avoided people | 0 | 1 | 2 | 3 | 9 |
| I tried to avoid meeting new people | 0 | 1 | 2 | 3 | 9 |

# Coping and in control

When you thought about your ostomy device and the risk of leakage, how did it affect your ability to cope?

| All of the time | Often | Sometimes | Rarely or never |
|---|---|---|---|
| 0 | 1 | 2 | 3 |
| 0 | 1 | 2 | 3 |
| 0 | 1 | 2 | 3 |
| 0 | 1 | 2 | 3 |
| | All of the time 0 0 0 0 | All of the time Often 0 1 0 1 0 1 0 1 | All of the time Often Sometimes 0 1 2 0 1 2 0 1 2 0 1 2 0 1 2 0 1 2 |

# 20.3. Appendix 3: Quality of life questionnaire

This questionnaire asks you about the use of the stoma appliance from this test period and your experiences. You will be asked questions about the discreetness of the stoma appliance, comfort relating to wearing the stoma appliance, confidence you have with the stoma appliance, and how the device impacts your social life.

Please think about your experience with using the stoma appliance **during the past seven days** and please select the box that is closest to your current situation. There are no right or wrong answers. We want to understand how beneficial you think the stoma appliance is and also what problems you may have experienced with it.

For each of the statements, think about how the specific issue affects you. Please answer **ALL** questions as honestly as you can, and **please remember to** answer the questions in relation to the past seven days only.

#### **HRQoL**

#### **Discreetness**

- 1. It was difficult to hide the stoma appliance under clothing
- 2. I was self-conscious about the appearance of the stoma appliance
- 3. The stoma appliance limited the choice of clothes that I could wear
- 4. The stoma appliance was obvious to other people
- 5. The color of the stoma appliance was discreet
- 6. It was difficult to hide the stoma appliance because of ballooning

#### Comfort

- 7. The stoma appliance was comfortable to wear
- 8. I was not concerned about skin irritation under the stoma appliance (for example, feelings of burning, itching, pinching or pain)
- 9. It was uncomfortable to remove the stoma appliance from my body
- 10. I often forgot that I was wearing the stoma appliance
- 11. The stoma appliance was comfortable as it fitted well to my body
- 12. The stoma appliance disrupted my sleep during the night

#### Confidence

- 13. I was confident that the stoma appliance would not leak
- 14. I worried that the stoma appliance would become loose from my body
- 15. I felt confident that I could spend the night away from home despite wearing the stoma appliance
- 16. I was confident the stoma appliance would not cause any problems for me
- 17. I felt confident to take part in physical activities (for example, sports) whilst wearing the stoma appliance
- 18. I worried that the stoma appliance would make a rustling noise.

#### Social life

- 19. I worried that my family and friends felt awkward around me because of the stoma appliance
- 20. I felt my social life had been restricted because of the stoma appliance
- 21. I avoided close physical contact with family and friends because of the stoma appliance
- 22. I worried about whether I could have a relationship because of my stoma appliance
- 23. I worried about whether the stoma appliance would affect my sex life

# 20.4. Appendix 4: Safety Interview guide

# Interview guide - Safety

# **Background information:**

The background information is asked to understand if the subject has experienced any problems or challenges during the test periods. And if so, in what situations and circumstances. The challenges can be changes in stoma behaviour, stoma shape, size or colour, abdominal troubles or changes in the subject general condition.

We will ask questions to understand when and why they have answered as they have to better understand how the test products differ from their own product.

- Introduce yourself
- Inform the subject about the purpose and background for the interview
- Use the following questions to lead the interview:
  - o How is your general health?
  - o How has your stoma behaved since your last visit?
  - o Has your stoma behaved differently since your last visit?
  - o How has your abdomen behaved since your last visit?
  - o Have you had any abdominal troubles?

# 20.5. Appendix 5: Interview guide (V6) and Follow-up

# Interview guide - V6 and follow-up

The following topics will be used as a guide during the interviews

- Introduction
- Experience throughout CP300
- Product change
- Their journey
- Products and routine
- Prototype review
- Close